CLINICAL TRIAL: NCT04083768
Title: Effect of Different Left Lateral Table Tilt on Neonatal Acid-base Status and Maternal Hemodynamics for Elective Cesarean Delivery Under Spinal Anesthesia
Brief Title: Effect of Different Left Lateral Table Tilt for Elective Cesarean Delivery Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Chao Xu, Principal Investigator, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XYFY2019-KL126-02
Record Dates: First submitted 2019-08-30; First posted 2019-09-10 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Elective Cesarean Section; Spinal Anesthesia
Keywords: Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supine group (Placebo Comparator): After the patient completes the spinal anesthesia, the cesarean section is completed in the supine position.
  Interventions: Device: 15° and 30° wedge sponges
- 15° group (Active Comparator): After the patient completed the spinal anesthesia, the preoperative preparation (about 10 minutes) was completed with a left tilt of 15°, and the cesarean section was completed using the supine position after the skin was cut.
  Interventions: Device: 15° and 30° wedge sponges
- 30° group (Active Comparator): After the patient completed the spinal anesthesia, the preoperative preparation (about 10 minutes) was completed with a left tilt of 30°, and the cesarean section was completed using the supine position after the skin was cut.
  Interventions: Device: 15° and 30° wedge sponges

INTERVENTIONS:
Device: 15° and 30° wedge sponges — After the spinal anesthesia is completed, the wedge sponge is placed between the patient's pelvis and ribs and the wedge is removed before the skin is cut.

SUMMARY:
The recommended position of the mother under caesarean section after spinal anesthesia is 15 degrees left. However, recent research has challenged the basic principles and practicality of the left-turn 15 degree position. Higuchi et al used nuclear magnetic imaging to directly prove that in the supine position, the position of the full-left 30 degrees of the full-term pregnancy of the full-term pregnancy relieved the inferior vena cava compression and the left-angle of 15 degrees did not. Therefore, there are more and more controversies about the choice of cesarean section position. This experiment aims to explore effects of different positions (15 degrees left, 30 degrees left and supine) for elective cesarean section on lumbar anesthesia for fetal acid-base balance and maternal Hemodynamic.

DETAILED DESCRIPTION:
When the pregnant woman in the third trimester is in the supine position, the enlarged uterus may oppress the inferior vena cava, thereby reducing the amount of blood and heart output of the pregnant woman. This affects the mother mainly, such as dizziness, nausea and vomiting, chills, and severe irritability，difficulty breathing or even cardiac arrest, the impact on the fetus is mainly the reduction of blood flow in the placenta, affecting the blood exchange of the uterus placenta, causing neonatal respiratory distress, acidosis and even death. The recommended position of the mother under caesarean section after spinal anesthesia is 15 degrees left. However, recent research has challenged the basic principles and practicality of the left-turn 15 degree position. Higuchi et al used nuclear magnetic imaging to directly prove that in the supine position, the position of the full-left 30 degrees of the full-term pregnancy of the full-term pregnancy relieved the inferior vena cava compression and the left-angle of 15 degrees did not. Therefore, there are more and more controversies about the choice of cesarean section position. This experiment aims to explore effects of different positions (15 degrees left, 30 degrees left and supine) for elective cesarean section on lumbar anesthesia for fetal acid-base balance and maternal Hemodynamic.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy at term via elective cesarean section
* Height from 150 cm to 180 cm
* American Society of Anesthesiologists (ASA) grade from I to II grade
* BMI（Body Mass Index，mearsured weight divided by height squared）less than 35 kg/m2.

Exclusion Criteria:

* Transverse lie
* Fetal macrosomia
* Uterine abnormalities (e.g., large fibroids, bicornuate uterus)
* Polyhydramnios
* Ruptured membranes
* Oligohydramnios
* Intrauterine growth restriction
* Gestational or nongestational hypertension, diabetes, eclampsia
* Hypertensive disorder or any condition associated with autonomic neuropathy (e.g., diabetes mellitus for more than 10 yr), with renal failure
* Have contraindications for spinal anesthesia（Such as low back infection, spinal deformity, etc.）
* Participants refused to sign informed consent.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Umbilical artery blood pH | Immediately after delivery
  Use a blood gas analyzer to measure

SECONDARY OUTCOMES:
Other UA and UV blood gas analysis values（pH, base excess, lactate , Umbilical artery blood PaCO2 | Immediately after delivery
  Use a blood gas analyzer to measure, PaCO2 in mmHg.
Fetal Apgar score (1 minute after birth) And 5 minutes | One minute and five minutes after the baby is delivered
  Measured by Apgar score.The Apgar scoring system is divided into five categories（muscle tone，heart rate，grimace and respiration) Appearance. Each category receives a score of 0 to 2 points. At most, a child will receive an overall score of 10（The higher the score, the better the child's condition）.
The incidence of nausea in pregnant women | Intraoperative
  Anesthesiologist observes combined patient dictation.
The incidence of vomiting in pregnant women | Intraoperative
  Anesthesiologist observes combined patient dictation
The incidence of hypotension in pregnant women | Intraoperative
  The increase of SBP <20% baseline SBP or SBP < 90/60mmHg
The incidence of hypertension in pregnant women | Intraoperative
  The increase of SBP >20% baseline SBP
The incidence of bradycardia in pregnant women | Intraoperative
  Heart rate less than 60 times per minute
One min (T1), 3 min (T2), 5 min (T3), 7 min (T4), 9 min (T5), 11 min (T6), 13 min (T7) and 15 min (T8) blood pressure after subarachnoid injection (completion of the subarachnoid injection was defined as 0 time point) | Intraoperative
  Measured by a sphygmomanometer.Systolic and diastolic blood pressure will be measured every minute during the study.
One min (T1), 3 min (T2), 5 min (T3), 7 min (T4), 9 min (T5), 11 min (T6), 13 min (T7) and 15 min (T8) heart rate after subarachnoid injection (completion of the subarachnoid injection was defined as 0 time point) | Intraoperative
  Obtained by ECG measurement
Dosage of phenylephrine during surgery | Intraoperative
  Used by an anesthesiologist based on the patient's blood pressure and heart rate.If the patient's blood pressure is less than 80% of the baseline level or less than 90/60 mmHg and the heart rate is greater than 60 times per minute, the patient is given 4 ug of phenylephrine.
Dosage of ephedrine during surgery | Intraoperative
  Used by an anesthesiologist based on the patient's blood pressure and heart rate.If the patient's blood pressure is less than 80% of the baseline level or less than 90/60 mmHg and the heart rate is smaller than 60 times per minute, the patient is given 6 mg of ephedrine.
Dosage of atropine during surgery | Intraoperative
  Used by an anesthesiologist based on the patient's blood pressure and heart rate.If the patient's heart rate is smaller than 60 times per minute, and blood pressure is more than 80% of the baseline level and more than 90/60 mmHg， the patient is given 0.5 mg of atropine.

CONTACTS AND LOCATIONS:
Locations (1):
- Liu Tian yu, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available when this trial is finished and the article have been published

REFERENCES:
- [Background] Fujita N, Higuchi H, Sakuma S, Takagi S, Latif MAHM, Ozaki M. Effect of Right-Lateral Versus Left-Lateral Tilt Position on Compression of the Inferior Vena Cava in Pregnant Women Determined by Magnetic Resonance Imaging. Anesth Analg. 2019 Jun;128(6):1217-1222. doi: 10.1213/ANE.0000000000004166. PMID 31094791
- [Background] Shayegan B, Khorasani A, Knezevic NN. Left Lateral Table Tilt for Elective Cesarean Delivery under Spinal Anesthesia Should Not Be Abandoned. Anesthesiology. 2018 Apr;128(4):860-861. doi: 10.1097/ALN.0000000000002095. No abstract available. PMID 29533301
- [Background] Abengochea A, Morales-Rosello J, Del Rio-Vellosillo M, Argente P, Barbera M. Effect of lateral tilt angle on the volume of the abdominal aorta and inferior vena cava in pregnant and nonpregnant women determined by magnetic resonance imaging. Anesthesiology. 2015 Sep;123(3):733-4. doi: 10.1097/ALN.0000000000000791. No abstract available. PMID 26284869
- [Result] Crawford JS, Burton M, Davies P. Time and lateral tilt at Caesarean section. Br J Anaesth. 1972 May;44(5):477-84. doi: 10.1093/bja/44.5.477. No abstract available. PMID 5044078
- [Derived] Liu T, Zou S, Guo L, Niu Z, Wang M, Xu C, Gao X, Shi Z, Guo X, Xiao H, Qi D. Effect of Different Positions During Surgical Preparation With Combined Spinal-Epidural Anesthesia for Elective Cesarean Delivery: A Randomized Controlled Trial. Anesth Analg. 2021 Nov 1;133(5):1235-1243. doi: 10.1213/ANE.0000000000005320. PMID 33350619